CLINICAL TRIAL: NCT05475587
Title: The Association Between Body Constitution and Meridian Energy Among Individuals With Prediabetes
Brief Title: The Association Between Body Constitution and Meridian Energy in Prediabetes
Status: Completed | Type: Observational
Sponsor: Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 07-XD-082
Record Dates: First submitted 2022-07-21; First posted 2022-07-27 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Prediabetes
Keywords: prediabetes; traditional Chinese medicine; body constitution
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prediabetes cases
  Interventions: Other: Routine care
- Healthy controls
  Interventions: Other: Routine care

INTERVENTIONS:
Other: Routine care — Both two groups received the same routine care.

SUMMARY:
Traditional Chinese medicine (TCM) theories assert that body constitution and meridian energy are the foundations for disease prevention. However, few studies have incorporated TCM concepts into risk factors. This study aimed to examine the association between body constitution and meridian energy in individuals with prediabetes. We conducted a matched case-control study that included 60 individuals with prediabetes. Finally, the reseachers have found that body constitution may be a risk factor fpr progression to type 2 diabetes mellitus in individuals with prediabetes.

DETAILED DESCRIPTION:
Objective: Traditional Chinese medicine (TCM) theories assert that body constitution and meridian energy are the foundations for disease prevention. However, few studies have incorporated TCM concepts into risk factors. This study aimed to examine the association between body constitution and meridian energy in patients with prediabetes.

Methods: The researchers conducted a matched case-control study from January to December 2019 that included 30 adults with prediabetes and 30 healthy controls, matched for age and sex, recruited from the outpatient clinic and health examination center at a teaching hospital in northern Taiwan. Body constitution was measured using the Body Constitution Questionnaire, which classifies the constitution as yang-deficiency, ying-deficiency, and phlegm-stasis, while meridian energy was measured using an Aetoscan meridian energy device (Aeto Technology Co. Ltd., Taiwan). The associations between body constitution, meridian energy, and prediabetes were examined using binary logistic regression analyses.

Conclusion: Body constitution may be a risk factor for progression to type 2 diabetes mellitus in patients with prediabetes and warrants further study.

ELIGIBILITY:
Inclusion Criteria:

* Previously diagnosed prediabetes with a hemoglobin A1c (HbA1c) of 5.7-6.4% and a f asting plasma glucose (FPG) of 100-125 mg/dL
* Aged ≥20
* provided informed consent
* The controls were healthy individuals whose FPG level was 100 mg/dL in at least two blood tests in the past 6 months.

Exclusion Criteria:

* Use of a hypoglycemic agent within the past 3 months
* Self-reported catastrophic illness in the last 6 months
* Pregnant and/or lactating
* Presence of pacemaker.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The researchers included 30 adults with prediabetes and 30 healthy controls, matched for age and sex, recruited from the outpatient clinic and health examination center at a teaching hospital in northern Taiwan.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Body constitution of body constitution questionnaire (BCQ) | One year
  The scale range from 44 to 220, with higher scores indicating larger deficiencies.

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Tzu Chi Hospital, New Taipei City, Taiwan